CLINICAL TRIAL: NCT05133895
Title: Pilot Study of Tocilizumab Monotherapy for Active Chronic Periaortitis
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Other Study IDs: Tocilizumab for Periaortitis
Record Dates: First submitted 2021-11-14; First posted 2021-11-24 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Chronic Periaortitis; Tocilizumab Monotherapy
Keywords: chronic periaortitis; Tocilizumab; treatment response; complete remission; partial remission
MeSH Terms: conditions — Retroperitoneal Fibrosis; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tocilizumab monotherapy: Patients with a definite or possible diagnosis of CP at acute active stage were enrolled for this study. Clinical diagnostic criteria consist of: (1) imaging findings show perivascular soft tissue density mass surrounding thoracic aorta, abdominal aorta or iliac arteries; (2) histopathological findings show fibrous tissue with chronic inflammatory infiltrate comprised of lymphocytes, plasma cells and macrophages (Neutrophils and granulomas are rare). Patients who satisfied (1) but without histopathological examination were perceived as possible CP. Secondary forms of CP related to drugs, infections, malignancies, Erdheim-Chester disease or other autoimmune diseases were excluded.
  Patients enrolled received intravenous infusions of TCZ (8 mg/kg) at inclusion and then every 4 weeks for at least 3 months.
  Interventions: Drug: Tocilizumab monotherapy

INTERVENTIONS:
Drug: Tocilizumab monotherapy — intravenous infusions of TCZ (8 mg/kg) at inclusion and then every 4 weeks for at least 3 months

SUMMARY:
This is a prospective study to investigate the treatment response of Tocilizumab on patients with active chronic periaortitis (CP).

Methods: patients with a definite or possible diagnosis of CP at acute active stage were enrolled for this study and accepted Tocilizumab monotherapy for 3 months.

Endpoints: The primary endpoint is to investigate the treatment response of Tocilizumab; the secondary endpoints include the improvement of inflammatory markers, the frequency of adverse events.

DETAILED DESCRIPTION:
Patients enrolled received intravenous infusions of TCZ (8 mg/kg) at inclusion and then every 4 weeks for at least 3 months. Demographic and clinical features, laboratory findings and imaging examinations were recorded at baseline and during 3-month follow-up. Imaging improvement was converted into the ratio of perivascular soft tissues shrinkage by evaluating 2 dimensions of greatest change on computed tomography (CT) at baseline and after 3 months. Partial remission was defined as obtaining alleviation of symptoms and normalization of inflammatory markers including erythrocyte sedimentation rate (ESR) and high-sensitivity C-reactive protein (hsCRP), with shrinkage of soft tissue mass in imaging <70%. Further, complete remission was defined as normalization of inflammatory markers accompanied by shrinkage of soft tissue mass ≥70%.

ELIGIBILITY:
Inclusion Criteria:

1. adults ≥ 18 years of age at time of informed consent;
2. meet clinical diagnostic criteria including (1) imaging findings show perivascular soft tissue density mass surrounding thoracic aorta, abdominal aorta or iliac arteries; (2) histopathological findings show fibrous tissue with chronic inflammatory infiltrate comprised of lymphocytes, plasma cells and macrophages (Neutrophils and granulomas are rare). Patients who satisfied (1) but without histopathological examination were perceived as possible CP;
3. at active stage: clinical symptoms or organ involvement; a higher level of ESR and CRP than normal;

Exclusion Criteria:

1. Secondary forms of CP related to drugs, infections, malignancies, Erdheim-Chester disease or other autoimmune diseases were excluded.
2. Combined with other autoimmune diseases.
3. Known immunodeficiency disorder.
4. Pregnancy, lactation, or planning to become pregnant within 6 months of the test.
5. Positive test for, or prior treatment for, hepatitis B or HIV infection. A positive test for hepatitis B is detection of hepatitis B surface antigen (HBsAg) or HBV-DNA.
6. Evidence of active tuberculosis (TB), including Chest X-ray and PPD.
7. Severe abnormal liver function or cardiac insufficiency.
8. Any reason the investigator think that should not attend this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic periaortitis (CP) is characterized by the presence of mass that develops around the thoracic aorta, abdominal aorta or iliac arteries, with predominance in males of middle and elderly age.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
treatment response | three months
  the rate of partial remission and complete remission after 3-month TCZ monotherapy

SECONDARY OUTCOMES:
the frequency of treatment related adverse events | three months
  adverse events caused by TCZ during 3-month follow-up.
the improvement of inflammatory markers | three months
  including erythrocyte sedimentation rate (ESR) and high-sensitivity C-reactive protein (hsCRP).

CONTACTS AND LOCATIONS:
Locations (1):
- Yunyun Fei, Beijing, China